CLINICAL TRIAL: NCT02633306
Title: Complex Oro-Facial Pain: Functional Imaging Characterization and Treatment With Transcranial Magnetic Stimulation
Brief Title: Transcranial Magnetic Stimulation for Facial Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1511M80284
Record Dates: First submitted 2015-12-10; First posted 2015-12-17 (Estimated); Results first posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-03

CONDITIONS: Trigeminal Nerve Injuries; Post-herpetic Neuralgia; Facial Pain; Nervus Intermedius Neuralgia
Keywords: trigeminal region pain
MeSH Terms: conditions — Trigeminal Nerve Injuries; Neuralgia, Postherpetic; Facial Pain; Myoclonic Cerebellar Dyssynergia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: This is a device study and therefore does not have a drug, biological/vaccine or combination product involved.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Transcranial Magnetic Stimulation (Experimental): transcranial magnetic stimulation
  Interventions: Device: transcranial magnetic stimulation

INTERVENTIONS:
Device: transcranial magnetic stimulation — Treatment will consist of five daily sessions of transcranial magnetic stimulation of the motor cortex contralateral to the pain.

SUMMARY:
Complex oro-facial pain is a poorly diagnosed and poorly treated cause of significant suffering and disability. This study will explore the ability of fMRI to identify patients with complex oro-facial pain who respond to transcranial magnetic stimulation therapy.

Specific Aims:

1. To establish baseline patterns of MRI in patients with chronic oro-facial pain without a definitive etiologic diagnosis.
2. To estimate the rate of treatment success of transcranial stimulation of the primary motor cortex (M1) in these patients.
3. To identify post-treatment MRI patterns that are associated with treatment success.

DETAILED DESCRIPTION:
Methods: Patients diagnosed with complex oral or facial pain at the UMPhysicians Complex Facial Pain Clinic who meet inclusion and exclusion criteria will be offered participation in the study. They will undergo baseline evaluation for depression with the HAM-D and MADRAS scales and for quality of life with the WHOQOL-BREF scale. Pain will be assessed using a 10 point visual analogue scale. Resting and pcasl MRI will be done within 24 hours before the first treatment. Treatment will consist of five daily sessions of motor cortex stimulation contralateral to the pain. Visual analogue pain scores will be obtained just before each treatment. Rating scales, resting and pcasl MRI will be repeated within 24 hours and at 2 weeks after the last treatment. Analysis: FMRI activation patterns will be examined by the investigators and correlated with treatment outcomes with the goal of identifying fMRI characteristics that can select patients suitable for further study.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 110
* Diagnosis of complex oro-facial pain made by the UMPhysicians Complex Facial Pain Clinic
* Alternative treatment of proven value not available as judged by the UMPhysicians Complex Facial Pain clinic
* One of the following types of facial pain as assessed by the Burchiel Patient Pain Rating Classification Questionnaire:

  * trigeminal neuralgia Type 2 (TN2)
  * trigeminal neuropathic pain (TNP)
  * trigeminal deafferentation pain (TDP)
  * post herpetic neuralgia (PHN)
  * atypical facial pain (AFP)
  * nervus intermedius neuralgia (NIN)
* Willing and able to give informed consent

Exclusion Criteria:

* Subject diagnosed according to the MINI as suffering from any other major Axis I disorder, such as Psychotic Disorder, Bipolar affective disorder, OCD (MDD is not contraindicated when Hamilton Depression Rating Scale -21≤26, or Beck Depression Inventory).
* Subjects with significant suicidal risk as assessed by the investigator using the Beck Suicide Ideation scale, psychiatric interview or a history of attempted suicide in the past year.
* Subject has a history of epilepsy or seizure (EXCEPT those therapeutically induced by ECT).
* Subject has a history of significant head trauma with loss of consciousness for longer than 5 minutes.
* Subject has a history of cranial surgery within 1 month of treatment.
* Subject has metallic particles in the eye or head (exclusive of mouth), implanted cardiac pacemaker or any intra-cardiac lines, implanted neurostimulators, intra-cranial implants (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or implanted medical pumps.
* Subject cannot pass the TMS Adult Safety Screen or the CMRR Safety Screen.
* Subject has severe and frequent headaches not part of their facial pain syndrome.
* Subject has a history of significant hearing loss.
* Subjects with a significant neurological disorder or insult including, but not limited to:

  * Any condition likely to be associated with increased intracranial pressure
  * Space occupying brain lesion
  * History of cerebrovascular accident
  * Transient ischemic attack within two years
  * Cerebral aneurysm
  * MMSE ≤ 24
  * Parkinson's disease
  * Huntington's chorea
  * Multiple sclerosis
* Subject with a history of substance abuse including alcoholism within the past 6 months (except nicotine and caffeine).
* Inadequate communication with the patient.
* Subject is under custodial care.
* Subject is currently participating in another clinical study or enrolled in another clinical study within 30 days prior to this study.
* Subject with unstable physical disease such as unstable cardiac disease.
* Subject is currently on Benzodiazepine at a dose higher than 3 mg of Lorazepam or equivalent.
* Subject has had previous treatment with TMS.
* Women who are breast-feeding.
* Women of childbearing potential and not using a medically accepted form of contraception when sexually active.
* Inability to give informed consent

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Haines, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Transcranial Magnetic Stimulation
Started | 9
Completed | 6
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: 2 of the 9 participants withdrew participant prior to the collection of baseline data. All 7 participants from whom data was collected are reported here.
Arm/Group | Transcranial Magnetic Stimulation
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 7
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Visual Analogue Scale (VAS)
Description: Participants are asked to rate pain on a100 mm visual analogue scale with 0 representing no pain and 100 representing worst possible pain. The mean difference from baseline to 7 days post-treatment is recorded.
Time Frame: 7 days
Population: Three patients left the study before treatment. One of 6 patients who began treatment did not complete the full treatment regimen and therefore post treatment status could not be assessed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transcranial Magnetic Stimulation
Number analyzed (Participants) | 5
score on a scale | 5.4 (11.7)
Statistical Analysis 1: Comparison: Transcranial Magnetic Stimulation; In an exploratory trial with such a small number of participants no statistical analysis beyond descriptive statistics of the findings is appropriate. The descriptive statistics are reported; Test type: Other; In an exploratory trial with such a small number of participants no statistical analysis beyond descriptive statistics of the findings is appropriate. The descriptive statistics are reported

2. Secondary Outcome: World Health Organization Quality of Life Abbreviated (WHOQOL-BREF) Overall
Description: A questionnaire used to determine the impact and burden of a disease on daily life. This assessment has 26 questions and covers the domains of physical and psychological health, social relationships, and environment. The answers to various question are included in one or more of the domains. Raw scores are transformed in several different ways by different investigators. We report raw scores. Domains have the following raw score ranges: Overall Quality of Life 2-10, Physical Heath 7-35, Psychological Health 6-30, Social Relationships 3-15, Environment 8-40, Total Raw Score 26-130. Higher scores in each of the domains correspond to greater perceived quality of life.
Time Frame: pre-treatment, 3 and 7 days post treatment
Population: All enrolled patients for whom any data was acquired are included.
Measure: Median (Full Range); unit: score on a scale
Groups:
- Transcranial Magnetic Stimulation: All patients enrolled 9 gave pretreatment data 6 gave 3 day post treatment data 5 gave 7 day post treatment data
  1 has missing data for 7 day post treatment social relationships score
Arm/Group | Transcranial Magnetic Stimulation
Number analyzed (Participants) | 9
score on a scale
  pre-treatment baseline | 5 [3 to 8]
  3 days post-treatment: number analyzed (Participants) | 6
  3 days post-treatment | 5 [4 to 8]
  7 days post-treatment: number analyzed (Participants) | 5
  7 days post-treatment | 5 [3 to 8]
Statistical Analysis 1: Comparison: Transcranial Magnetic Stimulation; [analysis description as in outcome 1, analysis 1]; Test type: Other; [other analysis details as in outcome 1, analysis 1]

3. Other Pre Specified Outcome: Young Mania Rating Scale (YMRS)
Description: The Young Mania Rating Scale (YMRS) is one of the most frequently utilized rating scales to assess manic symptoms. The scale has 11 items and is based on the patient's subjective report of his or her clinical condition over the previous 48 hours.
  The YMRS total score ranges from 0 to 60 where higher scores indicate more severe mania.
Time Frame: pre-treatment, 3 and 7 days post treatment
Population: all enrolled patients
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Transcranial Magnetic Stimulation
Number analyzed (Participants) | 9
score on a scale
  baseline | 0 [0 to 2]
  3 days post treatment: number analyzed (Participants) | 6
  3 days post treatment | 0 [0 to 1]
  7 days post treatment: number analyzed (Participants) | 5
  7 days post treatment | 0 [0 to 1]
Statistical Analysis 1: Comparison: Transcranial Magnetic Stimulation; [analysis description as in outcome 1, analysis 1]; Test type: Other; [other analysis details as in outcome 1, analysis 1]

4. Secondary Outcome: World Health Organization Quality of Life Abbreviated (WHOQOL-BREF) Physical Health
Description: as for outcome 2
Time Frame: baseline, 3 and 7 days post treatment
Population: All enrolled patients
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Transcranial Magnetic Stimulation
Number analyzed (Participants) | 9
score on a scale
  baseline | 19 [15 to 28]
  3 days post-treatment: number analyzed (Participants) | 6
  3 days post-treatment | 18.5 [15 to 21]
  7 days post-treatment: number analyzed (Participants) | 5
  7 days post-treatment | 17 [14 to 19]
Statistical Analysis 1: Comparison: Transcranial Magnetic Stimulation; [analysis description as in outcome 1, analysis 1]; Test type: Other; [other analysis details as in outcome 1, analysis 1]

5. Secondary Outcome: World Health Organization Quality of Life Abbreviated (WHOQOL-BREF) Psychological Health
Description: as for outcome 2
Time Frame: baseline, 3 and 7 days post treatment
Population: All enrolled patients
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Transcranial Magnetic Stimulation
Number analyzed (Participants) | 9
score on a scale
  baseline | 23 [17 to 28]
  3 days post-treatment: number analyzed (Participants) | 6
  3 days post-treatment | 22 [18 to 26]
  7 days post-treatment: number analyzed (Participants) | 5
  7 days post-treatment | 25 [12 to 27]
Statistical Analysis 1: Comparison: Transcranial Magnetic Stimulation; [analysis description as in outcome 1, analysis 1]; Test type: Other; [other analysis details as in outcome 1, analysis 1]

6. Secondary Outcome: World Health Organization Quality of Life Abbreviated (WHOQOL-BREF) Social Relationships
Description: as for outcome 2
Time Frame: baseline, 3 and 7 days post treatment
Population: All enrolled patients
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Transcranial Magnetic Stimulation
Number analyzed (Participants) | 9
score on a scale
  baseline | 13 [9 to 15]
  3 days post-treatment: number analyzed (Participants) | 6
  3 days post-treatment | 13 [9 to 15]
  7 days post-treatment: number analyzed (Participants) | 4
  7 days post-treatment | 13.5 [4 to 15]
Statistical Analysis 1: Comparison: Transcranial Magnetic Stimulation; [analysis description as in outcome 1, analysis 1]; Test type: Other; [other analysis details as in outcome 1, analysis 1]

7. Secondary Outcome: World Health Organization Quality of Life Abbreviated (WHOQOL-BREF) Environment
Description: as for outcome 2
Time Frame: baseline, 3 and 7 days post treatment
Population: All enrolled patients
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Transcranial Magnetic Stimulation
Number analyzed (Participants) | 9
score on a scale
  baseline | 37 [24 to 40]
  3 days post-treatment: number analyzed (Participants) | 6
  3 days post-treatment | 37 [31 to 39]
  7 days post-treatment: number analyzed (Participants) | 5
  7 days post-treatment | 38 [32 to 43]
Statistical Analysis 1: Comparison: Transcranial Magnetic Stimulation; [analysis description as in outcome 1, analysis 1]; Test type: Other; [other analysis details as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Transcranial Magnetic Stimulation
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transcranial Magnetic Stimulation (N=6)
Increased Pain (General disorders) | 1 (1)
Tremors (Nervous system disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Headache (General disorders) | 1 (1)
Non-specific Pain (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2021-01-21): https://cdn.clinicaltrials.gov/large-docs/06/NCT02633306/Prot_000.pdf